CLINICAL TRIAL: NCT05168878
Title: Safety Education in the Emergency Department (SEED): A Pilot Study
Brief Title: Safety Education in the Emergency Department: A Pilot Study
Acronym: SEED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado Clinical & Translational Sciences Institute (Other); Emergency Medicine Foundation (Other); American Foundation for Firearm Injury Reduction in Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-0238; CMH-M-20-15 (Other Grant/Funding Number: Colorado Clinical and Translational Sciences Institute)
Record Dates: First submitted 2021-11-23; First posted 2021-12-23 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-08

CONDITIONS: Firearm Injury
Keywords: Injury prevention; anticipatory guidance; firearm counseling

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patient > 9 yo, no video (No Intervention): Caregivers of patients greater than or equal to 10 years old will not be shown a video in the PED.
- Patient > 9 yo, 3 minute video (Active Comparator): Caregivers of patients greater than or equal to 10 years old will be shown a 3-minute BeSMART video in the PED.
  Interventions: Behavioral: 3-minute BeSMART video
- Any age, 30-second video (Experimental): Caregivers of patients of any age will be shown a 30 second BeSMART video in the PED.
  Interventions: Behavioral: 30-second BeSMART video
- Any age, 3 minute video (Experimental): Caregivers of patients of any age will be shown a 3-minute BeSMART video in the PED.
  Interventions: Behavioral: 3-minute BeSMART video

INTERVENTIONS:
Behavioral: 30-second BeSMART video — 30 second video focused on education about child gun deaths and responsible gun storage
  Arms: Any age, 30-second video
Behavioral: 3-minute BeSMART video — 3-minute video focused on education about child gun deaths and responsible gun storage
  Arms: Any age, 3 minute video; Patient > 9 yo, 3 minute video

SUMMARY:
The purpose of this pilot study is to assess the feasibility and acceptability of video-based safe firearm storage education in the Pediatric Emergency Department.

ELIGIBILITY:
Inclusion criteria:

* Children > 30 days and < 18 years old presenting to the CHCO ED
* Parent/guardian who is ≥ 18 and ≤ 85 years old
* Arms 1 & 2 will include a subset of patients ≥10 years and < 18 years old with a firearm in the home.

Exclusion criteria:

* Child is in an emergent/acute medical condition
* Patient seen in our fast track area or other room without a television
* Parent/guardian is non-English speaking.

Ages: 30 Days to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 407 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maya Haasz, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

REFERENCES:
- [Derived] Haasz M, Betz ME, Ambroggio L, Cafferty R, King CA, Wong S, Leonard J, Brooks-Russell A, Sigel E. Acceptability and feasibility of video-based firearm safety education in a Colorado emergency department for caregivers of adolescents in firearm-owning households. Inj Prev. 2026 Jan 20;32(1):90-97. doi: 10.1136/ip-2023-045204. PMID 39053924

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patient > 9 yo, no Video | Patient > 9 yo, 3 Minute Video | Any Age, 30-second Video | Any Age, 3 Minute Video
Started | 95 | 62 | 127 | 123
Completed | 51 | 23 | 45 | 46
Not Completed | 44 | 39 | 82 | 77

BASELINE CHARACTERISTICS:
Groups:
- Patient > 9 yo, 3-minute Video: Caregivers of patients greater than or equal to 10 years old will be shown a 3-minute BeSMART video in the PED.
  3-minute BeSMART video: 3-minute video focused on education about child gun deaths and responsible gun storage
- Any Age, 30-second Video: Caregivers of patients of any age will be shown a 30-second BeSMART video in the PED.
  30-second BeSMART video: 30-second video focused on education about child gun deaths and responsible gun storage
- Any Age, 3-minute Video: Caregivers of patients of any age will be shown a 3-minute BeSMART video in the PED.
  3-minute BeSMART video: 3-minute video focused on education about child gun deaths and responsible gun storage
- Total: Total of all reporting groups
Arm/Group | Patient > 9 yo, no Video | Patient > 9 yo, 3-minute Video | Any Age, 30-second Video | Any Age, 3-minute Video | Total
Number analyzed (Participants) | 95 | 62 | 127 | 123 | 407
Age, Customized [Count of Participants; unit: Participants]
  Age: <24 | 0 | 0 | 8 | 8 | 16
  Age: 25-34 | 11 | 8 | 51 | 41 | 111
  Age: 35-44 | 47 | 31 | 48 | 58 | 184
  Age: 45-54 | 36 | 19 | 12 | 14 | 81
  Age: >55 | 1 | 4 | 8 | 2 | 15
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 77 | 56 | 106 | 100 | 339
  Gender: Male | 18 | 4 | 20 | 21 | 63
  Gender: Unknown | 0 | 2 | 1 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 14 | 32 | 42 | 106
  Not Hispanic or Latino | 73 | 44 | 85 | 72 | 274
  Unknown or Not Reported | 4 | 4 | 10 | 9 | 27

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Intervention
Description: Acceptability of the educational videos measured using agreement with the question, "Overall I liked the video". Responses will be on a Likert scale with 1 being the lowest and 5 being the highest.
Time Frame: At baseline
Population: All basline participants
Measure: Count of Participants; unit: Participants
Arm/Group | Patient > 9 yo, 3 Minute Video | Any Age, 30-second Video | Any Age, 3 Minute Video
Number analyzed (Participants) | 62 | 127 | 123
Participants
  Overall liked the video (agree/ strongly agree) | 49 | 104 | 109
  Overall liked the video (Neutral/ disagree/ strongly disagree) | 13 | 23 | 14

2. Primary Outcome: Feasibility of Follow up
Description: Feasibility of completing a follow up survey with parents within 3 months after the intervention measured by the proportion of caregivers who complete the survey in its entirety either electronically or by phone.
Time Frame: Through study completion, an average of three months
Measure: Count of Participants; unit: Participants
Arm/Group | Patient > 9 yo, no Video | Patient > 9 yo, 3 Minute Video | Any Age, 30-second Video | Any Age, 3 Minute Video
Number analyzed (Participants) | 95 | 62 | 127 | 123
Participants
  Followed up at three months | 51 | 23 | 45 | 46
  Did not follow up at three months | 44 | 39 | 82 | 77

3. Primary Outcome: Safe Firearm Storage
Description: Self- report based on the survey question, "Are any of the guns in your home kept unlocked?" at baseline. This question has a yes/ no answer.
Time Frame: At baseline
Population: Any guns kept unlocked at baseline. Only recorded for patient>9 years old as these patients were all firearm owners whereas "all ages" group had both firearm owners and non-firearm owners.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient > 9 yo, no Video | Patient > 9 yo, 3 Minute Video
Number analyzed (Participants) | 95 | 62
Participants
  Are any of the guns in your home kept unlocked? - yes at baseline | 9 | 5
  Are any of the guns in your home kept unlocked? - no at baseline | 86 | 57

4. Primary Outcome: Safe Firearm Storage at Three Months
Description: Self- report at two time points based on the survey question, "Are any of the guns in your home kept unlocked?" at three month follow up; yes/ no answer.
Time Frame: Three month follow up
Population: Any guns kept unlocked at follow up. Only analyzed for arms of study where all caregivers are firearm owners.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient > 9 yo, no Video | Patient > 9 yo, 3 Minute Video
Number analyzed (Participants) | 47 | 18
Participants
  Are any of the guns in your home kept unlocked? - yes at follow-up | 7 | 0
  Are any of the guns in your home kept unlocked? - no at follow-up | 40 | 18

5. Primary Outcome: Knowledge About Temporary Firearm Transfer at Baseline
Description: Parental awareness of temporary firearm transfer will be measured by self-report based on question, "Did you know that you can temporarily take your guns out of your home if you are concerned that someone in your house may hurt themselves or someone else?". (responses answers are yes or no) OR ability to name at least one location for temporary firearm storage OR describe the link for a map of storage locations.
Time Frame: At baseline
Population: Knowledge of temporary transfer at baseline
Measure: Count of Participants; unit: Participants
Groups:
- Patient All Ages, 30-second Video: Caregivers of patients shown 30-second video
- Patient All Ages, 3-minute Video: Caregivers of patients shown 3-minute video
Arm/Group | Patient > 9 yo, no Video | Patient > 9 yo, 3 Minute Video | Patient All Ages, 30-second Video | Patient All Ages, 3-minute Video
Number analyzed (Participants) | 95 | 62 | 127 | 123
Participants
  Knowledge of temporary transfer at baseline - Yes | 69 | 47 | 28 | 33
  Knowledge of temporary transfer at baseline - No | 26 | 15 | 99 | 90

6. Primary Outcome: Knowledge About Temporary Firearm Transfer at Follow up
Description: Parental awareness of temporary firearm transfer will be measured by self-report based on question, "Did you know that you can temporarily take your guns out of your home if you are concerned that someone in your house may hurt themselves or someone else?". (responses answers are yes or no) and ability to name at least one location for temporary firearm storage OR describe the link for a map of storage locations.
Time Frame: At study follow-up, an average of three months
Population: Number of participants who answered the question and reported knowledge of temporary transfer of firearms out of the home at 3 month follow up.
Measure: Count of Participants; unit: Participants
Groups:
- Patient > 9 yo, no Video: Caregivers of patients greater than or equal to 10 years old will not be shown a video in the PED. Follow up
- Patient > 9 yo, 3 Minute Video: Caregivers of patients greater than or equal to 10 years old will be shown a 3-minute BeSMART video in the PED.
  3-minute BeSMART video: 3-minute video focused on education about child gun deaths and responsible gun storage. Follow up
- Patient All Ages, 30-second Video: Caregivers of patients shown 30-second video. Follow up
- Patient All Ages, 3-minute Video: Caregivers of patients shown 3-minute video. Follow up.
Arm/Group | Patient > 9 yo, no Video | Patient > 9 yo, 3 Minute Video | Patient All Ages, 30-second Video | Patient All Ages, 3-minute Video
Number analyzed (Participants) | 49 | 19 | 13 | 16
Participants | 44 | 18 | 13 | 14

ADVERSE EVENTS:
Time Frame: Three months
Description: The plan was for any adverse events to be reported directly to the PI.
Arm/Group | Patient > 9 yo, no Video | Patient > 9 yo, 3 Minute Video | Any Age, 30-second Video | Any Age, 3 Minute Video
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/62 | 0/127 | 0/123
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/62 | 0/127 | 0/123
Other Adverse Events (participants affected / at risk) | 0/95 | 0/62 | 0/127 | 0/123

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-17): https://cdn.clinicaltrials.gov/large-docs/78/NCT05168878/Prot_SAP_000.pdf